CLINICAL TRIAL: NCT05557045
Title: Phase 1, FIH, Open-label, Nonrandomized, Multicenter Study of JZP815 in Participants With Advanced or Metastatic Solid Tumors Harboring Alterations in the MAPK Pathway
Brief Title: A Study of JZP815 Oral Capsules in Adult Participants With Advanced or Metastatic Solid Tumors Harboring Mitogen Activated Protein Kinase (MAPK) Pathway Alterations to Investigate the Safety, Dosing, and Antitumor Activity of JZP815
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JZP815-101
Record Dates: First submitted 2022-09-12; First posted 2022-09-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Advanced Cancer; Metastatic Cancer; Solid Tumor
Keywords: Advanced Cancer; Metastatic Cancer; Solid Tumor; JZP815
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Exploration (Part A): JZP815 (Experimental): Participants will receive JZP815 with a starting dose of 20 mg twice daily (BID).
  Interventions: Drug: JZP815
- Expansion (Part B): JZP815 (Experimental): Participants with advanced or metastatic solid tumors who will receive JZP815 at the RP2D established in Dose Exploration (Part A).
  Interventions: Drug: JZP815

INTERVENTIONS:
Drug: JZP815 — JZP815 will be administered as oral capsules to participants BID approximately 12 hours apart, in the morning and in the evening. QD dosing may also be investigated, if supported by PK data.

SUMMARY:
This phase 1 study will investigate the safety, dosing, and initial antitumor activity of JZP815 in participants with advanced or metastatic solid tumors harboring alterations in the MAPK pathway.

DETAILED DESCRIPTION:
This first-in-human study will consist of two parts: Part A and Part B.

Part A will characterize the safety and tolerability of JZP815, assess pharmacokinetics (PK) profile, and determine a recommended phase 2 dose (RP2D) to be further investigated in the Expansion phase (Part B).

Part B will further investigate the RP2D determined in Part A, and assess antitumor activity in various subsets of disease (based on mutation and/or tumor type) in which the mechanism of action of JZP815 is applicable.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age, at the time of signing the informed consent
* Participants who have histological or cytological diagnosis of an advanced or metastatic solid tumor carrying a documented, clinically significant, MAPK pathway alteration
* Participants must have exhausted all available standard of care therapies, or in the opinion of the investigator would be unlikely to tolerate or derive clinically meaningful benefit from available standard of care therapy
* Performance status (ECOG) of 0 or 1, measured within 72 hours before start of treatment. For Arm 7 (NRAS Q61 mutated anaplastic thyroid cancer) in Part B (Expansion), ECOG of 0 to 2, measured within 72 hours before the start of treatment.
* Must have measurable disease by RECIST v1.1
* Tumor must be safely amenable to core needle or excisional biopsy (applies only to participants enrolled in Pre-Expansion cohorts)
* Adequate organ function
* Expected life expectancy of at least 12 weeks
* For each arm in Part B (Expansion), participants must be diagnosed with the tumor type(s) carrying the mutation(s) specified and meet protocol specified requirements for prior therapy
* Male participants must agree to refrain from donating sperm plus either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or must agree to use contraception
* Female participants are eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: is a women of nonchildbearing potential (WONCBP) or is a women of childbearing potential (WOCBP) and using a contraceptive method that is highly effective during the study intervention period and for at least 3 months after the last dose of study intervention and agrees not to donate eggs
* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum) within 3 days before the first dose of study intervention
* Capable of giving signed informed consent

Exclusion Criteria:

* Known uncontrolled brain metastases. Stable brain metastases either treated or being treated with a stable dose of steroids/anticonvulsants, with no dose change in the previous 4 weeks, are permitted
* Active fungal, bacterial and/or known viral infection including HIV or Hepatitis A, B, C
* Concomitant malignancies or previous malignancies with less than 2 years disease-free interval at the time of enrollment, with the exception of non-metastatic, non-melanomatous skin cancers, carcinoma in-situ, melanoma in-situ, prostate cancer with undetectable PSA, indolent thyroid cancer that are adequately treated
* Has clinically significant (ie, active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (> New York Heart Association Classification Class II), QTc ≥ 470 msec, or serious cardiac arrhythmia requiring medication
* Uncontrolled or severe intercurrent medical condition
* Gastrointestinal condition that could impair absorption of study intervention or inability to ingest study intervention
* In the judgement of the investigator, any important medical illness or abnormal laboratory finding that would increase the risk of participating in this study
* Received any cancer directed therapy (chemotherapy, hormonal therapy, biologic, etc.) within 28 days or 5 half-lives (whichever is shorter) of starting study intervention. For Arm 7 (NRAS Q61 mutated anaplastic thyroid cancer) in Part B (Expansion), participants who have received radio-sensitizing chemotherapy (low-dose chemotherapy) are permitted a wash-out period of 7 days or 5 half-lives, whichever is shorter (a discussion with the sponsor is required). Participants who have received radiotherapy must have recovered from acute toxicities associated with treatment.
* Use of any products or medicines known to be strong or moderate inducers or inhibitors of CYP3A4, which cannot be discontinued at least 4 weeks or 5 half-lives (whichever is shorter) before starting study intervention, or planned use at any time during the study
* Use of proton pump inhibitors (eg, omeprazole) and histamine-2 receptor antagonists (eg, famotidine), which cannot be discontinued at least 2 weeks before first dose, or planned use at any time during the study
* Concurrent therapy with any other investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose-Limiting Toxicities (Part A) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Number of Participants With Treatment-emergent Adverse Events and Serious Adverse Events (Part A and B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Change From Baseline in Hemoglobin (Part A and B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Change From Baseline in Absolute Neutrophil Count (Part A and B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Change From Baseline in Platelets (Part A and B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Change From Baseline in Hematocrit (Part A and B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Change From Baseline in Aspartate Aminotransferase (Part A and B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Change From Baseline in Alanine Aminotransferase (Part A and B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Change From Baseline in Creatinine (Part A and B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Change From Baseline in Total Bilirubin (Part A and B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Change From Baseline in Heart Rate (Part A and B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Change From Baseline in Blood Pressure (Part A and B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Number of Participants With Dose Interruptions and Reductions (Part A and B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Objective Response Rate (as Defined by RECIST v1.1) (Part B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Duration of Response (Part B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention

SECONDARY OUTCOMES:
Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) Levels of JZP815 and its Metabolites (Part A) | MTD determination cohorts, Cycle 1 Days 1 and 15: predose and 0.25,0.5,1,2,3,4,6, 8 hours (hr) postdose; 24, 48 and 72 hr postdose relative to 1st dose given on Cycle 1 Day 1; Others, Cycle 1 Days 1, 15 or 22: predose and 0.25,0.5,1,2,3,4,6,8 hr postdose
Pharmacokinetic Parameter Time to Maximum Plasma Concentration (Tmax) of JZP815 and its Metabolites (Part A) | MTD determination cohorts, Cycle 1 Days 1 and 15: predose and 0.25,0.5,1,2,3,4,6, 8 hours (hr) postdose; 24, 48 and 72 hr postdose relative to 1st dose given on Cycle 1 Day 1; Others, Cycle 1 Days 1, 15 or 22: predose and 0.25,0.5,1,2,3,4,6,8 hr postdose
Pharmacokinetic Parameter Area Under the Concentration-Time Curve (AUC) of JZP815 and its Metabolites (Part A) | MTD determination cohorts, Cycle 1 Days 1 and 15: predose and 0.25,0.5,1,2,3,4,6, 8 hours (hr) postdose; 24, 48 and 72 hr postdose relative to 1st dose given on Cycle 1 Day 1; Others, Cycle 1 Days 1, 15 or 22: predose and 0.25,0.5,1,2,3,4,6,8 hr postdose
  AUC from time 0 to infinity (AUCinf) and AUC during a dosing interval (AUCtau) will be assessed.
Pharmacokinetic Parameter Apparent Terminal Elimination Half-life (t1/2) of JZP815 and its Metabolites (Part A) | MTD determination cohorts, Cycle 1 Days 1 and 15: predose and 0.25,0.5,1,2,3,4,6, 8 hours (hr) postdose; 24, 48 and 72 hr postdose relative to 1st dose given on Cycle 1 Day 1; Others, Cycle 1 Days 1, 15 or 22: predose and 0.25,0.5,1,2,3,4,6,8 hr postdose
Pharmacokinetic Parameter Clearance (CL/F) of JZP815 (Part A) | MTD determination cohorts, Cycle 1 Days 1 and 15: predose and 0.25,0.5,1,2,3,4,6, 8 hours (hr) postdose; 24, 48 and 72 hr postdose relative to 1st dose given on Cycle 1 Day 1; Others, Cycle 1 Days 1, 15 or 22: predose and 0.25,0.5,1,2,3,4,6,8 hr postdose
Pharmacokinetic Parameter Accumulation Ratio of JZP815 and its Metabolites (Part A) | MTD determination cohorts, Cycle 1 Days 1 and 15: predose and 0.25,0.5,1,2,3,4,6, 8 hours (hr) postdose; 24, 48 and 72 hr postdose relative to 1st dose given on Cycle 1 Day 1; Others, Cycle 1 Days 1, 15 or 22: predose and 0.25,0.5,1,2,3,4,6,8 hr postdose
Pharmacokinetic Parameter Apparent Volume of Distribution During Terminal Phase (Vz/F) of JZP815 (Part A) | MTD determination cohorts, Cycle 1 Days 1 and 15: predose and 0.25,0.5,1,2,3,4,6, 8 hours (hr) postdose; 24, 48 and 72 hr postdose relative to 1st dose given on Cycle 1 Day 1; Others, Cycle 1 Days 1, 15 or 22: predose and 0.25,0.5,1,2,3,4,6,8 hr postdose
Pharmacokinetic Parameter Metabolite to Parent Ratio of JZP815 and its Metabolites (Part A) | MTD determination cohorts, Cycle 1 Days 1 and 15: predose and 0.25,0.5,1,2,3,4,6, 8 hours (hr) postdose; 24, 48 and 72 hr postdose relative to 1st dose given on Cycle 1 Day 1; Others, Cycle 1 Days 1, 15 or 22: predose and 0.25,0.5,1,2,3,4,6,8 hr postdose
Objective Response Rate (as Defined by RECIST v1.1) (Part A) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Progression-free Survival (Part B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention
Overall Survival (Part B) | Baseline until death, withdrawal of consent, or lost to follow-up, up to 18 months after last participant starts study intervention

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - SCRI HealthOne, Denver, Colorado
  - Florida Cancer Specialists - Lake Nona, Orlando, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - University of Chicago, Chicago, Illinois
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Oklahoma University, Oklahoma City, Oklahoma
  - Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - Texas Oncology- Central South, Austin, Texas
  - Texas Oncology- Gulf Coast, The Woodlands, Texas
  - Virginica Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No